CLINICAL TRIAL: NCT04456556
Title: Combined Endophthalmitis and Orbital Cellulitis in Patients With Novel Coronavirus Disease (COVID-19)
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Farouk Sayed Othman Abelkader, associate professor, Minia University
Other Study IDs: ocular infection in covid19
Record Dates: First submitted 2020-06-30; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Endophthalmitis and Orbital Cellulitis
Keywords: endophthalmitis; orbital cellulitis; covid-19
MeSH Terms: conditions — Endophthalmitis; Orbital Cellulitis; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To report on cases presented with combined endophthalmitis and orbital cellulitis as a first presentation of covid-19 infection.

DETAILED DESCRIPTION:
This observation case series study included 5 patients referred to the Ophthalmology Department, Minia University with severe ophthalmic manifestations in the form of combined endophthalmitis and orbital cellulitis. On doing the work-up of covid-19 infection according to the recommendations of Egyptian Ministry of Health, patients proved to be infected by the novel Corona virus. In addition to the Corona work-up, all patients were subjected to full ophthalmological evaluation, ocular ultrasound and orbital CT examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with endophthalmitis and orbital cellulitis with covid-19

Exclusion Criteria:

* Patients without endophthalmitis and orbital cellulitis.
* Patients with endophthalmitis and orbital cellulitis not having covid-19 infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 5 patients referred to the Ophthalmology Department, Minia University with severe ophthalmic manifestations in the form of combined endophthalmitis and orbital cellulitis. On doing the work-up of covid-19 infection according to the recommendations of Egyptian Ministry of Health, patients proved to be infected by the novel Corona virus.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Combined Endophthalmitis and Orbital Cellulitis in patients with Novel Coronavirus Disease (COVID-19) | baseline
  highlight the occurrence of combined endophthalmitis and orbital cellulitis in patients with novel Coronavirus Disease (COVID-19)

CONTACTS AND LOCATIONS:
Locations (1):
- Minia university Hospital, Minya, Minya Governorate, Egypt

REFERENCES:
- [Background] Chen L, Liu M, Zhang Z, Qiao K, Huang T, Chen M, Xin N, Huang Z, Liu L, Zhang G, Wang J. Ocular manifestations of a hospitalised patient with confirmed 2019 novel coronavirus disease. Br J Ophthalmol. 2020 Jun;104(6):748-751. doi: 10.1136/bjophthalmol-2020-316304. Epub 2020 Apr 7. PMID 32265202
- [Background] Turbin RE, Wawrzusin PJ, Sakla NM, Traba CM, Wong KG, Mirani N, Eloy JA, Nimchinsky EA. Orbital cellulitis, sinusitis and intracranial abnormalities in two adolescents with COVID-19. Orbit. 2020 Aug;39(4):305-310. doi: 10.1080/01676830.2020.1768560. Epub 2020 May 18. PMID 32419568
- [Background] Elshafei AMK, Sayed MF, Abdallah RMA. Clinical profile and outcomes of management of orbital cellulitis in Upper Egypt. J Ophthalmic Inflamm Infect. 2017 Dec;7(1):8. doi: 10.1186/s12348-017-0126-3. Epub 2017 Mar 9. PMID 28275981
- [Derived] Abdelkader MFSO, Elshafei AMK, Nassar MM, Abu Elela MA, Abdallah RMA. Combined endophthalmitis and orbital cellulitis in patients with corona virus disease (COVID-19). J Ophthalmic Inflamm Infect. 2021 Sep 15;11(1):27. doi: 10.1186/s12348-021-00258-y. PMID 34523045